CLINICAL TRIAL: NCT05503784
Title: Study to Evaluate the Efficacy of Bite's Natural Deodorant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kind Lab PBC. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20227
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Sweat; Underarm Odor
Keywords: sweat; underarm odor; perspiration

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bite Deodorant (Experimental): All 38 participants apply BITE deodorant daily for four weeks.
  Interventions: Other: BITE Deodorant

INTERVENTIONS:
Other: BITE Deodorant — BITE natural Deodorant

SUMMARY:
This is an open-label observational single-arm clinical trial to study the efficacy of a commercial deodorant and its effect on odor, clothing (stains), and quality of life. It is hypothesized that the deodorant marketed as Bite deodorant will mask bodily odor in participants, will not stain clothes, and improve the quality of life in trial participants.

ELIGIBILITY:
Inclusion Criteria:

* Agree to refrain from the use of any other deodorant or antiperspirant other than Bite for the study period
* Must be in good health (does not report any medical conditions asked in the screening questionnaire)
* Must be willing to comply with the requirements of the protocol
* Must be willing to add the deodorant to their daily routine
* Is willing and able to share feedback
* Shower daily, and put deodorant on the first thing in the morning (before sweating)
* If used deodorants previously must be a natural version

Exclusion Criteria:

* Unwilling to follow the routine of the protocol
* Currently participating in another research study
* Severe chronic conditions including oncological conditions, psychiatric disease, or other
* Females that are pregnant, want to become pregnant for the duration of the study, or who are breastfeeding
* Presence of self-reported armpit sensitivity
* Known to have severe allergic reactions
* Have known allergies to the trial product ingredients
* Currently using an antiperspirant

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in underarm odor | 4 weeks
  Survey-based assessment (0-5 scale) of changes in underarm odor
Changes in clothing staining | 4 weeks
  survey-based assessment (0-5 scale) of changes in clothing staining
Changes in reported quality of life | 4 weeks
  survey-based assessment (0-5 scale) of changes in reported quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided